CLINICAL TRIAL: NCT02885259
Title: Subcutaneous Immunoglobulin With rHuPH20 in Multifocal Motor Neuropathy
Brief Title: HyQvia in Multifocal Motor Neuropathy
Acronym: HYMMNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, L.H. van den Berg, Professor dr, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL52642.041.15
Record Dates: First submitted 2016-01-25; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Multifocal Motor Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HyQvia (Experimental): human immunoglobulin and one vial of recombinant human hyaluronidase (rHuPH20
  Interventions: Drug: rHuPH20

INTERVENTIONS:
Drug: rHuPH20 — human immunoglobulin and one vial of recombinant human hyaluronidase
  Other Names: HyQvia

SUMMARY:
Subcutaneous immunoglobulin (SCIG) and recombinant human hyaluronidase (rHuPH20) will be tested in patient witch MMN and currently under maintenance treatment with IVIG for safety, tolerability and efficacy.

DETAILED DESCRIPTION:
Multifocal motor neuropathy (MMN) is a chronic immune mediated neuropathy, which affects patients at a relatively young age and necessitates treatment with immunoglobulins (Ig) to improve and maintain muscle strength. Subcutaneous immunoglobulin (SCIG) therapy for MMN is equally efficacious to intravenous immunoglobulin (IVIG), may be self-administered and may induce fewer systemic adverse reactions. However, limited subcutaneous infusion volumes and reduced bioavailability, necessitate multiple infusion sites, more frequent treatment, and dose adjustment to achieve pharmacokinetic equivalence. This is an issue in particular in MMN where relatively high and frequent doses are necessary to maintain long-term improvement of muscle strength. Recombinant human hyaluronidase (rHuPH20) increases subcutaneous tissue permeability and facilitates dispersion and absorption, enabling subcutaneous administration of higher (monthly) doses of Ig. If treatment with HyQvia is at least equally effective and safe as compared with conventional Ig treatment, HyQvia could become the preferred treatment option for patients with MMN as it may have attractive benefits for patients by its mode of administration.

Objective:

The primary objective is to study the safety and tolerability of HyQvia in patients with

MMN as compared with conventional intravenous, by documenting:

* Side effects by using a diary and a 10 cm visual analogue scale (VAS) scales to measure headache and nausea.
* Biochemical tests (Hemoglobin, haptoglobin, reticulocyte counts, lactate dehydrogenase, bilirubin, DAT) for haemolytic anemia 3-7 days after the last IVIG/SCIG infusion, during the enrolment period and 3-7 days after the last HyQvia infusion during the treatment period.
* Anti- hyaluronidase antibody titer before and after/during the HyQvia treatment. Together with the above mentioned test parameters in point 2, each time 30ml (equal to three tubes) will be drawn.
* Patient satisfaction of product on a 10 cm VAS scale.

The secondary objective is to determine the efficacy of treatment with HyQvia in patients with MMN on:

* Disability, measured by Guy's Neurological Disability Scale and the self-evaluation scale;
* Function, measured by a nine hole peg test (9-HPT) and a 40 meter walk test (40-MWT);
* Muscle strength, measured by manual muscle testing and hand-held dynamometry.

Study design:

HyQvia in MMN will be studied in a prospective, uncontrolled single-blind open-label study of 20 patients on IVIG with a duration of 48 to 60 weeks consisting of:

1. Enrolment period of 12 to 24 weeks' duration in which patients will be treated according to their regular maintenance treatment regimen with IVIG, and visit the outpatient clinic every 6 weeks.
2. Treatment period of 9 months' duration in which patients will be treated with HyQvia, using the same dose as during the enrolment period and visit the outpatient clinic at start and after 6, 12, 24 and 36 weeks.
3. During the study, the dose may be increased if patients' functioning in daily life is worsening: the score of either the upper or lower limb score of the Guy's Neurological Disability Scale or the score of at least two motor activities on the self- evaluation scale have increased with 1 point or muscle strength on hand-held dynamometry has worsened by 50% or more in at least two clinically affected muscles or muscle groups. If patients do not improve on increased Ig dose during the treatment period the investigator can decide to stop maintenance treatment with HyQvia and restart the previous treatment after a period of minimal 3 months.

HyQvia will be administrated in patients' routine setting -at home or in the hospital- with help of a nurse who is trained in using HyQvia. The patients are carefully monitored for potential adverse signs throughout the study period as well as anti- hyaluronidase antibody induction.

Study population:

From the outpatient clinic at the UMC Utrecht, 20 patients with MMN and currently under maintenance treatment with IVIG will be selected to study the safety, tolerability and efficacy of HyQvia.

Intervention: 20 MMN patients, currently under maintenance treatment with IVIG, will be will be treated with HyQvia during a 9 months' period using the same dose as IVIG during the enrolment period.

Main study parameters/endpoints:

The following main study parameters will be used to assess tolerability and efficacy of HyQvia in MMN patients:

* Disability using the Guy's Neurologic Disability Scale and the self- evaluation scale.
* Function will be evaluated with a 9-HPT and a 40 MWT.
* Muscle strength will be measured with manual muscle testing using the Medical Research Council scale (MRC). Hand-held dynamometry will be performed in a selection of those muscles or muscle groups with an MRC score < 5 at any time. Grip strength of the hands will be measured using a hand-held dynamometer.
* Adverse events by using 10 cm long VAS analogue scales for headache and nausea as well as a diary, which will be provided to the patient at each visit in the clinic.
* IgM anti-GM1 ganglioside antibody titers at the enrolment visit and at the final visit.

Biochemical tests for haemolytic anemia 3-7 days after the last IVIG/SCIG infusion during the enrolment period and 3-7 days after the last HyQvia infusion during the treatment period.

* Anti-hyaluronidase antibody titer 12 weeks before and at 3 and 9 months during HyQvia treatment. Together with the above mentioned test parameters in point 5, each time 30ml (equal to three tubes) will be drawn.
* Patient satisfaction of product on a 10 cm VAS scale.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The risks are negligible and the burden minimal for patients enrolled in this study, assessing tolerability and efficacy of HyQvia in MMN patients. Patients participating in the study, will be assigned 6 grouped evaluations at fixed intervals: filling out a diary, evaluation scales, 3 blood samples, visit the outpatient clinic and are also evaluated with routine physical examinations. The two components of HyQvia, Subcutaneous immunoglobulin (SCIG) and recombinant human hyaluronidase (rHuPH20), are known to be safe and are already applied in primary and secondary immunodeficiency disorders, multiple myeloma and chronic lymphatic leukemia. SCIG therapy for MMN, is safe and equally efficacious to intravenous immunoglobulin (IVIG). Furthermore, it may be self-administered and may induce fewer systemic adverse reactions than IVIG. Recombinant human hyaluronidase (rHuPH20), increases subcutaneous tissue absorption and enables higher doses of subcutaneous administration Ig, which will decrease the number of infusion sites, resulting in less frequent treatment and dose adjustments.

ELIGIBILITY:
Inclusion Criteria:

1. Age at onset of MMN, 18 - 99 years.
2. The presence of asymmetrical limb weakness at onset or motor involvement having a motor nerve distribution in at least two peripheral nerve distributions, predominant upper limb involvement, disabling weakness MRC grade 4 or less in at least one muscle.
3. Decreased or absent tendon reflexes in affected limbs.
4. Electrophysiological evidence of one site with definite motor conduction block or one site with probable conduction block according to previously defined criteria.
5. Response to IVIG according to criteria that were described in previous studies.
6. Stable on IVIG maintenance treatment in the year preceding the study.
7. Patients have given written informed consent, prior to the study, with the understanding that consent may be withdrawn at any time without prejudice.

Exclusion Criteria:

1. Bulbar signs or symptoms.
2. Upper motor neuron signs (spasticity, hyperreflexia, extensor plantar response).
3. Sensory symptoms and signs with sensory deficits on examination (except for vibration sense) and abnormal results of sensory nerve conduction studies
4. Other neuropathies (e.g. diabetic, lead, porphyric or vasculitic neuropathy, chronic inflammatory demyelinating polyneuropathy, Lyme neuroborreliosis, post radiation neuropathy, hereditary neuropathy with liability to pressure palsies, Charcot-Marie-Tooth neuropathies, meningeal carcinomatosis).
5. Treatment with other immunosuppressive drugs (cyclophosphamide, azathioprine, cyclosporin) in the 6 months preceding the study.
6. Female patient who is pregnant or breast-feeding or of childbearing potential.

   Confirmation that the patient is not pregnant will be established by a negative b-HCG test within a 7-day period before inclusion in the study. Lack of childbearing potential is met by:
   1. being post-menopausal,
   2. being surgically sterile,
   3. practising contraception with an oral contraceptive, intra-uterine device, diaphragm or condom with spermicide or d) being sexually inactive.
7. Age < 18 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured by anamnesis | 1 year
  presence of headache, gastrointestinal complaints, fatigue, flue-like symptoms

SECONDARY OUTCOMES:
Quality of life (QoL) measured by a VAS questionnaire | 1 year
  VAS questionnaire every visit at the outpatient clinic.
Stability of muscle strength | 1 year
  Every visit at the outpatient clinic a Guy's neurologic disability scale (GNDS) and MRC sum score are obtained
Safety measured by questionnaire | 1 year
  QoL questionnaire measured in a VAS number
Safety measured by blood test | 1 year
  Liver tests and blood counts

CONTACTS AND LOCATIONS:
Overall Officials: Leonard van den Berg, prof, Principal Investigator — UMCU
Locations (1):
- UMCU, Utrecht, Utrechts, Netherlands

IPD SHARING:
Plan to Share IPD: No